CLINICAL TRIAL: NCT01099995
Title: Phase 3 Study of Hyperbaric Oxygen Therapy for Comatose Patients With Acute Domestic Carbon Monoxide Poisoning
Brief Title: Hyperbaric Oxygen Therapy for Comatose Patients With Acute Carbon Monoxide Poisoning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the study was halted after the first interim analysis as there were significantly more patients who recovered at one month in the control arm
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Misse, DRRC AP-HP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO89-2
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Carbon Monoxide Poisoning
Keywords: domestic accident; coma; carbon monoxide; intoxication; acute domestic carbon monoxide poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning; Coma | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One HBO session (Active Comparator): hyperbaric oxygen therapy one dive at 2 absolute atmosphere (1-hour plateau) - oxygen was delivered via a full face mask - followed by 4 hours of normobaric oxygen therapy
  Interventions: Other: Hyperbaric oxygen therapy
- 2 HBO sessions (Experimental): Two sessions of hyperbaric oxygen therapy at 2 absolute atmosphere (1-hour plateau) with oxygen delivered via a full face mask at 100% inspired oxygen fraction or via mechanical ventilation
  Interventions: Other: hyperbaric oxygen therapy

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — one dive at 2 absolute atmosphere (1-hour plateau) with 30 min time for compression and decompression - oxygen was delivered via a full face mask at high concentration to achieve a 100% inspired fraction of oxygen or via mechanical ventilation
  Arms: One HBO session
Other: hyperbaric oxygen therapy — two dives at 2 absolute atmosphere (1-hour plateau) with 30 min of compression and 30 min of decompression - oxygen being delivered via a full face mask at 100% inspired oxygen fraction or via mechanical ventilation
  Arms: 2 HBO sessions

SUMMARY:
Carbon monoxide poisoning still places a burden on the healthcare system worldwide. While oxygen therapy is the cornerstone treatment, the role and practical modalities of hyperbaric oxygen therapy (HBO) remain controversial. This study aimed at comparing two sessions of HBO at 2 absolute atmosphere and one session of HBO at 2 absolute atmosphere followed by 4 hours of normobaric oxygen therapy in comatose adult victims of acute domestic carbon monoxide poisoning.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 15 years of age
* admitted for domestic CO poisoning within 12 hours after the end of CO exposure
* initial coma, regardless of consciousness at hospital admission
* carboxyhemoglobin level at presentation greater than 10% or 5%, in smokers and non-smokers, respectively

Exclusion Criteria:

* poisoning by more than one compound (e.g., CO plus a drug or CO plus other toxic gases such as those found in fire smoke)
* suicide attempt
* pregnancy
* contraindications to HBO (circulatory collapse or pneumothorax)
* technical obstacles to HBO
* non domestic CO poisoning
* difficulty in determining whether the patient experienced initial loss of consciousness or initial coma
* consent refusal

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1989-10; Primary Completion 2000-01 (Actual); Study Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
complete recovery | at one month
  Complete recovery was defined as an absence of symptoms reported on the self-assessment questionnaire with a normal physical exam (including normal neuropsychological functions).

SECONDARY OUTCOMES:
persistent neurological sequels | at one month
  Neurological sequels were considered persistent (PNS) if they were present both at hospital discharge and at one-month evaluation, regardless of the type of manifestation.
delayed neurological sequels | at one month
  Delayed neurological sequelae (DNS) were any neurological manifestations that appeared between hospital discharge and one-month evaluation, regardless of their severity. Patients with DNS were those considered fully recovered at hospital discharge but with neurological manifestations at one-month evaluation.
the difference in carboxyhemoglobin levels before/after treatment completion | at 12 hours from randomization
  the difference between serum levels of carboxyhemoglobin at baseline and those recorded immedaitely after study treatment completion
serious adverse events | at one month
  any complication of hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, Study Chair — Assistance Publique - Hôpitaux de Paris; Jean Claude Raphael, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Raymond Poincaré Hospital, Garches, France